CLINICAL TRIAL: NCT04967248
Title: Alpelisib (Piqray®) Post-Authorization Safety Study (PASS): a Non-interventional Study of Alpelisib in Combination With Fulvestrant in Postmenopausal Women, and Men, With Hormone Receptor Positive (HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-), Locally Advanced or Metastatic Breast Cancer With a Phosphatidylinositol-3-kinase Catalytic Subunit Alpha (PIK3CA) Mutation, After Disease Progression Following Endocrine Therapy as Monotherapy, in the Real-world Setting
Brief Title: A NIS of Alpelisib in Combination With Fulvestrant in Postmenopausal Women, and Men, With HR+,HER2- , Locally Advanced or Metastatic Breast Cancer With a PIK3CA Mutation, After Disease Progression Following Endocrine Therapy as Monotherapy, in the Real-world Setting
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719C2404
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Hormone Receptor Positive HER2 Negative Breast Cancer With a PIK3CA Mutation
Keywords: Breast Cancer; non-interventional study; NIS; alpelisib; fulvestrant; PASS
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- alpelisib in combination with fulvestrant: Patients treated with alpelisib in combination with fulvestrant
  Interventions: Other: Alpelisib; Other: Fulvestrant

INTERVENTIONS:
Other: Alpelisib — Prospective observational PASS study. There was no treatment allocation. Patients recruited on or before their first prescribed dose of alpelisib in combination with fulvestrant were enrolled.
Other: Fulvestrant — Prospective observational PASS study. There was no treatment allocation. Patients recruited on or before their first prescribed dose of alpelisib in combination with fulvestrant were enrolled.

SUMMARY:
This was a prospective, multi-national, non-interventional study (NIS) collecting data from postmenopausal women, and adult men, with HR+, HER2- locally advanced or metastatic breast cancer whose tumor harbors a PIK3CA mutation, and who were to be treated with alpelisib in combination with fulvestrant after disease progression following endocrine therapy as monotherapy, in the real-world setting.

DETAILED DESCRIPTION:
Once the patient provided informed consent, he or she was enrolled in the study. Patients were planned to be followed from enrollment until 1) 30 days after alpelisib treatment discontinuation, or 2) death, or 3) lost to follow-up, or 4) patient withdrawal, or 5) physician decision to end treatment/study, or 6) end of the study, whichever occured first. The end of the study was defined as a maximum of 12 months after the date the last patient was enrolled (LPFV); if the last patient was still on treatment on that date, they were not be followed up any further.

Due to very low patient numbers (4 patients, including 2 eligible patients) no statistical analyses were performed. Database lock was achieved without all queries resolved.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from the patient or a legally acceptable representative, obtained before any study-related activities are undertaken
* Patients diagnosed with HR+, HER2- locally advanced or metastatic breast cancer with a PIK3CA mutation
* Patients who have disease progression following endocrine therapy as monotherapy
* Patients must be postmenopausal women, or men, ≥18 years of age
* Patients recruited on or before their first prescribed dose of alpelisib in combination with fulvestrant

Exclusion Criteria:

* Use of alpelisib prior to signing the informed consent form for this study
* Participation in an interventional study within 30 days prior to the initiation of alpelisib

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women, and adult men, with HR+, HER2- locally advanced or metastatic breast cancer whose tumor harbors a PIK3CA mutation, and who were treated with alpelisib in combination with fulvestrant after disease progression following endocrine therapy as monotherapy, in the real-world setting.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Incidence proportion of hyperglycemia | Up to 53 months
  To assess the incidence of hyperglycemia (Adverse Event of Special Iinterest) observed during follow-up of patients treated with alpelisib in combination with fulvestrant.

SECONDARY OUTCOMES:
Calculated BMI | Baseline
  Calculated BMI will be collected
Medical history | Baseline
  Number of patients with diabetes mellitus (including gestational diabetes), tobacco use, baseline diabetic status per laboratory values for HbA1c and FPG
Family history of diabetes mellitus | Baseline
  Yes/ No variable
Number of patients with concomitant medications known to affect blood glucose levels | Baseline
  Number of patients with concomitant medications known to affect blood glucose levels will be measured
Number of participants with incidence proportion of ketoacidosis and Hyperglycemic Hyperosmolar Non-Ketotic Syndrome (HHNKS) | Up to 53 months
  Number of participants with incidence proportion of ketoacidosis and HHNKS based on AE data
Incidence of the Adverse Events of Special Interest (AESI) of Osteonecrosis of the Jaw (ONJ) | Up to 53 months
  Incidence of AESI of Osteonecrosis of the Jaw (ONJ) will be provided
Number of participants with risk factors for Osteonecrosis of the Jaw (ONJ) observed | Baseline
  Number of participants with risk factors for ONJ will be collected. Risk factors for ONJ include:
  * Patient characteristics: age, calculated BMI, sex
  * Prior and/or concomitant use of bisphosphonates (e.g. zoledronic acid).
  * Prior and/or concomitant use of RANKligand inhibitors (e.g. denosumab).
Incidence proportion of AESIs | Up to 53 months
  The incidence proportion of AESIs:
  * GI toxicity (nausea, vomiting and diarrhea)
  * Rash
  * Hypersensitivity (e.g. anaphylactic reaction)
  * Pancreatitis
  * Pneumonitis
  * SCARs
Other safety and tolerability events | Up to 53 months
  The incidence proportion of:
  * AEs
  * AEs leading to dose interruptions
  * AEs leading to dose reductions
  * AEs leading to permanent discontinuation of alpelisib in combination with fulvestrant
  * SAEs
Number of patients with hematological and biochemical laboratory abnormalities | Up to 53 months
  Number of patients with hematological and biochemical laboratory abnormalities will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18363